CLINICAL TRIAL: NCT06849492
Title: An Open, Multicenter Study on the Treatment of Recurrent and Metastatic Triple-negative Breast Cancer Guided by Cell Surface Protein Typing (HIM) in Triple-negative Breast Cancer
Brief Title: HIM Typing Guides the Treatment of Advanced First-Line Triple-Negative Breast Cancer
Acronym: SHIFT-001
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Chief physician, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHIFT-001
Record Dates: First submitted 2025-02-16; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Advanced Triple Negative Breast Cancer
MeSH Terms: interventions — camrelizumab; 130-nm albumin-bound paclitaxel; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A (H subtyping) (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Nab-paclitaxel
- Cohort B (I subtyping) (Experimental)
  Interventions: Drug: SKB264
- Cohort C (M subtyping) (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Nab-paclitaxel; Drug: Lenvatinib

INTERVENTIONS:
Drug: Camrelizumab — PD-1 inhibitor
  Arms: Cohort A (H subtyping); Cohort C (M subtyping)
Drug: Nab-paclitaxel — chemotherapy
  Arms: Cohort A (H subtyping); Cohort C (M subtyping)
Drug: SKB264 — Trop2-ADC
  Arms: Cohort B (I subtyping)
Drug: Lenvatinib — Anti-angiogenic TKI
  Arms: Cohort C (M subtyping)

SUMMARY:
To explore the efficacy and safety of treatment for recurrent and metastatic advanced first-line triple-negative breast cancer guided by cell surface protein-based subtyping (HIM).

ELIGIBILITY:
Inclusion Criteria:

1. More than 18 years old;
2. ECOG PS Score: 0~1;
3. Patients must have a life expectancy ≥ 3 months;
4. Histopathologically confirmed recurrent metastatic triple-negative invasive breast cancer (HER2-negative: IHC 0/1+ or IHC 2+ with negative ISH; ER-negative: IHC <1%, PR-negative: IHC <1%)；
5. At least one measurable lesion according to RECIST 1.1 criteria；
6. No prior systemic anti-tumor therapy during the recurrent or metastatic stage；
7. Sufficient tissue samples for HIM subtyping analysis (at least 15 unstained slides from the most recent metastatic lesion biopsy are required; primary lesion samples from treatment-naive patients are acceptable, and re-biopsy samples from such patients are also acceptable)；
8. Adequate organ function and marrow function;
9. Willing to join in this study, able to provide written informed consent, good compliance and willing to cooperate with follow-up.

Exclusion Criteria:

1. Has leptomeningeal metastasis or cystic metastatic lesions confirmed by MRI or lumbar puncture;
2. Existence of third space fluid (e.g. massive ascites, pleural effusion, pericardial effusion) that is not well controlled by effective methods, e.g.；
3. Received systemic anti-tumor therapy within 14 days prior to enrollment;
4. Imaging shows tumor invasion of major blood vessels, or the investigator judges that the tumor is highly likely to invade critical vessels during the study period, leading to life-threatening hemorrhage；
5. Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, serum calcium > 12 mg/dL, or albumin-corrected serum calcium > ULN); or symptomatic hypercalcemia requiring ongoing bisphosphonate therapy；
6. Prior treatment with immune checkpoint inhibitors other than PD-1/PD-L1 monoclonal antibodies (including but not limited to CTLA-4 antibodies, etc.), or anti-angiogenic agents (including monoclonal antibodies and TKIs)；
7. History of other malignancies within the past 5 years, having received any systemic anti-tumor therapy or local treatment (including surgery and radiotherapy) for malignancies, excluding cured in situ carcinomas, cervical carcinoma, basal cell carcinoma, squamous cell carcinoma, thyroid carcinoma, and other malignancies;
8. Major surgery unrelated to breast cancer within 4 weeks prior to enrollment, or the patient has not fully recovered from such surgical procedures (tissue biopsy for diagnostic purposes and peripherally inserted central catheter placement are allowed);
9. Any known or suspected autoimmune disease, except for: hypothyroidism due to autoimmune thyroiditis requiring only hormone replacement therapy; or stable type I diabetes with controlled blood glucose;
10. Presence of interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, pulmonary fibrosis, acute pneumonia, etc.);
11. History of live or attenuated live vaccination within 28 days prior to the first study dose or planned live or attenuated live vaccination during the study period;
12. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); active hepatitis (hepatitis B, defined as HBV-DNA ≥ 30 copies/ml; hepatitis C, defined as HCV-RNA above the lower limit of detection of the assay method) or co-infection with hepatitis B and C; autoimmune hepatitis;
13. Severe infections within 4 weeks prior to the first dose, including but not limited to bacteremia or severe pneumonia requiring hospitalization; or active infections requiring systemic antibiotic treatment with CTCAE ≥ grade 2 within 2 weeks prior to the first dose; or unexplained fever > 38.5°C during screening or prior to the first dose (fever due to tumor-related causes, as judged by the investigator, is allowed); evidence of active tuberculosis infection within 1 year prior to dosing;
14. History of or planned allogeneic bone marrow transplantation or solid organ transplantation;
15. Peripheral neuropathy ≥ grade 2;
16. Severe cardiac disease or conditions；
17. Subjects who have received systemic immunostimulant therapy (including but not limited to interferon or interleukin-2, including immunostimulants in clinical research stages) within 4 weeks prior to the first dose;
18. Subjects who have received systemic immunosuppressive therapy (including but not limited to glucocorticoids, azathioprine, methotrexate, thalidomide, anti-tumor factor drugs) within 2 weeks prior to the first dose. This exclusion does not apply to intranasal and inhaled corticosteroids or physiological doses of systemic steroid hormones (i.e., no more than 10 mg/day prednisone or equivalent doses of other corticosteroids)；
19. Known allergy to the investigational drug or any of its excipients; or a history of severe allergic reactions to other monoclonal antibodies;
20. Female patients during the gestation or suckling period, of childbearing potential and pregnancy test-positive, or unwilling to use an effective method of contraception during the whole study;
21. A documented history of neurological or psychiatric disorders, including epilepsy or dementia, or a known history of substance abuse, alcoholism, or drug addiction.
22. Any other conditions not appropriate for study enrolment in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | at the time point of every 12 weeks, up to one year
  ORR is the percentage of evaluable patients with a confirmed investigator-assessed target lesion response of CR (complete response) or PR (partial response) per RECIST 1.1

SECONDARY OUTCOMES:
CBR | up to 2 years
  CBR is the percentage of evaluable patients with a confirmed investigator-assessed target lesion response of CR (complete response) or PR (partial response) or at least 6 months of SD (stable disease) per RECIST 1.1
DoR | up to 2 years
  DoR is the time from the date of first detection of objective response (which is subsequently confirmed) until the date of objective radiographic disease progression.
PFS | up to 2 years
  PFS is the time from the date of first dose until the date of objective radiographic disease progression or death (by any cause in the absence of progression).
OS | up to 3 years
  OS is the time from the date of first dose until the date of death by any cause.
Safety | from time of informed consent provided to 3 months after the last dose of study therapy
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Percentage of participants who experienced an adverse event and discontinued study drug due to an AE.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No